CLINICAL TRIAL: NCT01774305
Title: Effect of Single-dose Dexmedetomidine on Airway Reflex in Adult With Oral Intubation After Thyroidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong Soo Lee, Yonsei university college of medicine, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2012-0142
Record Dates: First submitted 2012-12-22; First posted 2013-01-23 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Coughing
MeSH Terms: conditions — Cough | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- dexmedetomidine (Experimental): We administrate the dexmedetomidine single bolus (0.5ug/kg, intravenously, for 10 min) at time of muscle layer closing.
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator): We administrate the saline single bolus (0.25ml/kg,intravenously, for 10 min) at time of muscle layer closing.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — We administrate the dexmedetomidine single bolus (0.5ug/kg, intravenously) at time of muscle layer closing.
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: Saline — We administrate the normal saline (single bolus, 0.25ml/kg) intravenously at time of muscle layer closing.
  Other Names: Normal saline
  Arms: saline

SUMMARY:
Coughing during emergence from general anaesthesia may lead to dangerous effects including laryngospasm, detrimental haemodynamic changes. Post-thyroidectomy bleeding occurs in 1-4% of patients, and severe coughing may cause bleeding. Dexmedetomidine, a potent α adrenoreceptor agonist, is theoretically appropriate for reducing airway and haemodynamic reflexes during emergence from anaesthesia.

In this study, we investigated whether intravenous single-dose dexmedetomidine at the end of surgery reduces coughing during extubation after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2 patients patients scheduled for thyroidectomy

Exclusion Criteria:

* Severe cardiovascular disease history of motion sickness active status of upper respiratory infection allergy to dexmedetomidine patients who cannot understand Korean

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JS, Choi SH, Kang YR, Kim Y, Shim YH. Efficacy of a single dose of dexmedetomidine for cough suppression during anesthetic emergence: a randomized controlled trial. Can J Anaesth. 2015 Apr;62(4):392-8. doi: 10.1007/s12630-014-0295-6. Epub 2014 Dec 19. PMID 25523837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period : Sep.2012. ~ Jan. 2013 types of location : medical clinic.
Pre-assignment Details: there was no specific pre-assignment details.
Period: Overall Study
Arm/Group | Dexmedetomidine | Saline
Started | 71 | 71
Completed | 70 | 71
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: A patient in group Dexmedetomidine was not completed this study due to changed surgery plan. (Intubated time prolonged more than 3 hours)
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Saline | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 71 | 141
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.4) | 45.6 (12.3) | 45.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 53 | 112
  Male | 11 | 18 | 29
smoking [Number; unit: participants] — It has been known that smoking history is related to coughing.
  participants
    smoking | 12 | 18 | 30
    non-smoking | 58 | 53 | 111

OUTCOME MEASURES:

1. Primary Outcome: Coughing Grade
Description: The coughing incidence and severity will be measured at extubation. Especially from the time of eye opening to 5 min after extubation. The coughing grade was assessed by the following cough grading system: Grade 0, no cough or single, mild cough at extubation; Grade 1, multiple, not sustained cough with mild severity; Grade 2, cough persistence less than 5 s with moderate severity; Grade 3, severe, persistent cough for more than 5 s (bucking).
Time Frame: from the time of eye opening to 5 min after extubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Saline
Number analyzed (Participants) | 70 | 71
units on a scale | 0.6 (0.9) | 1.4 (0.9)

2. Secondary Outcome: Emergence Time
Description: The emergence time will be recorded as the time from sevoflurane discontinuation to eye opening on command.
Time Frame: from sevoflurane discontinuation, up to the time of eye opening (estimated time : from 5 min to 10 min)
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Dexmedetomidine | Saline
Number analyzed (Participants) | 70 | 71
sec | 492 (176) | 355 (151)

ADVERSE EVENTS:
Time Frame: 3 hours
Description: prolonged intubation more than 3 hrs, due to changed surgical plan.
Arm/Group | Dexmedetomidine | Saline
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 1/71 | 0/71
OTHER ADVERSE EVENTS (reported when occurring in more than 1.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=71) | Saline (N=71)
prolonged intubation (Surgical and medical procedures) | 1 (1) | 0 (0) — 1 patient in Dex group was intubated more than 3 hrs due to changed surgical plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No